CLINICAL TRIAL: NCT02559050
Title: Nasal Reconstruction Using a Customized 3D-printed Nasal Stent for Congenital Arhinia
Status: Completed | Type: Observational
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Pohang University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jong-Won Rhie MD.PhD, Professor, Seoul St. Mary's Hospital
Other Study IDs: SM-AR-01
Record Dates: First submitted 2015-08-26; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Arhinia
MeSH Terms: conditions — Arrhinia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Customized 3D-printed nasal stent — Silicone stent with unconventional shape, 3D-printed based on patient's computed topographical images, to exactly fit newly made nasal cavity.

SUMMARY:
A 7-year-old arhinia patient receives nasal reconstruction with nasal cavity reconstruction and is aided with the application of a 3D-printed nasal stent to prevent nasal cavity constriction.

DETAILED DESCRIPTION:
After reconstruction of a nasal cavity in the maxilla by burring using a navigation system, the patient required a nasal stent to prevent stenosis. However there was no conventional stent available. A 3D-printed silicone nasal stent was custom made for the cavity and inserted.

ELIGIBILITY:
Inclusion Criteria:

* Single patient
* 7-year-old male
* Congenital arhinia
* No history of previous treatment

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A 7-year-old male patient with congenital arhinia with no history of previous treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Nasal cavity diameter | 6 months
  Change from baseline nasal cavity diameter (measured by CT sagittal section, in millimeters)

REFERENCES:
- [Derived] Jung JW, Ha DH, Kim BY, Seo BF, Han HH, Kim DH, Rhie JW, Kim SW, Cho DW. Nasal Reconstruction Using a Customized Three-Dimensional-Printed Stent for Congenital Arhinia: Three-Year Follow-up. Laryngoscope. 2019 Mar;129(3):582-585. doi: 10.1002/lary.27335. Epub 2018 Sep 24. PMID 30247752